CLINICAL TRIAL: NCT05096143
Title: A Cohort Study to Compare the Hospitalization Between Naive Sacubitril/Valsartan and Naive ACEi/ARBs Heart Failure Patients With Reduced Ejection Fraction Using Secondary US Electronic Health Records Data
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696B2036
Record Dates: First submitted 2021-10-19; First posted 2021-10-27 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
Keywords: Heart failure hospitalizations,; sacubitril/valsartan,; Angiotensin II receptor antagonist,; United States,; electronic health record
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Naive Sacubitril/valsartan: Participants who were prescribed with Naive Sacubitril/valsartan
  Interventions: Drug: Sacubitril/valsartan
- Naive ACEi/ARB: Participants who were prescribed with Naive Angiotensin-converting enzyme inhibitors/Angiotensin II receptor antagonists (ACEi/ARB)
  Interventions: Drug: ACEi/ARB

INTERVENTIONS:
Drug: Sacubitril/valsartan — Participants who were prescribed with Sacubitril/valsartan
  Other Names: Entresto®
  Groups: Naive Sacubitril/valsartan
Drug: ACEi/ARB — Participants who were prescribed with Angiotensin-converting enzyme inhibitors/Angiotensin II receptor antagonists (ACEi/ARB)
  Groups: Naive ACEi/ARB

SUMMARY:
A non-interventional retrospective cohort study conducted to compare the naive sacubitril/valsartan Heart Failure with reduced Ejection Fraction (HFrEF) patient population to a matched naive ACEi/ARB HFrEF patient population.

DETAILED DESCRIPTION:
This was a non-interventional retrospective cohort study using the US secondary EHR dataset, Optum EHR, to compare the naive sacubitril/valsartan HFrEF patient population (aged ≥ 18 years) to a matched naive ACEi/ARB HFrEF patient population.

The study comprised of the following periods:

Identification period: 01-Jul-2015 to 31-Mar-2019

Study period

* 01-Jul-2014 to 31-Mar-2020 for primary objective and secondary objective 2 to 6.
* 01-Jul-2008 to 30-Sep-2020 for secondary objective 1.

Follow-up period: Patients were followed up until 31-Mar-2020, death or patient transfer out.

Baseline period: 365 days prior to index

ELIGIBILITY:
Inclusion Criteria:

Sacubitril/valsartan incident cohort Included patients

* Prescribed sacubitril/valsartan within the identification period (01-July-2015 to 31-Mar-2019), that had non-missing gender and year of birth data.
* With at least one ICD-9-CM or ICD-10-CM code for diagnosis of HF within one-year prior to date of first prescription of sacubitril/valsartan (index date), and are treated as part of the integrated delivery network.
* With first month active 365 days prior to index and last date active was greater than or equal to (≥) index, and the month of provider source data was greater than the final date of patient follow-up.
* That were ≥18 years old at index date.
* With a valid LVEF value ≤40%, prior to index (index date included).

Angiotensin-converting enzyme inhibitors (ACEi) and Angiotensin II receptor antagonist (ARB) incident cohort

Included patient:

* Prescribed ACEi or ARBs within the identification period (01-Jul-2015 to 31-Mar-2019), that had non-missing gender and year of birth data.
* With at least one ICD-9-CM or ICD-10-CM code for diagnosis of HF within one-year prior to date of first prescription of ACEi or ARB (index date), and were treated as part of the integrated delivery network.
* With first month active 365 days prior to index and last date active was ≥ index, and the month of provider source data is greater than the final date of patient follow-up.
* That were ≥ 18 years old at index date.
* With a valid LVEF value ≤ 40%, prior to index (index date included).

Exclusion Criteria:

Sacubitril/valsartan incident cohort

Excluded patients for the primary objective and secondary objective 2 to 6:

* Patients who were prescribed sacubitril/valsartan within one-year prior to index date.
* Patients who were prescribed ACEi or ARBs, within one-year prior to index date (index date included).

Exclude patients for secondary objective 1:

* Patients who were prescribed sacubitril/valsartan prior to index date.
* Patients who were prescribed ACEi or ARBs prior to index date (index date included).

Angiotensin-converting enzyme inhibitors (ACEi) and Angiotensin II receptor antagonist (ARB) incident cohort

Exclude patients for the primary objective and secondary objective 2 to 6:

* Patients who were prescribed ACEi or ARBs within one-year prior to index date.
* Patients who were prescribed sacubitril/valsartan within one-year prior to index date (index date included).
* Which had a valid sacubitril/valsartan prescription that enables inclusion in the sacubitril/valsartan cohort.
* Exclude patients for secondary objective 1:
* Patients who were prescribed ACEi or ARBs prior to index date.
* Patients who were prescribed sacubitril/valsartan prior to index date (index date included).
* Which had a valid sacubitril/valsartan prescription that enables inclusion in the sacubitril/valsartan cohort

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included heart failure patients with reduced ejection fraction
Sampling Method: Probability Sample
Enrollment: 42269 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Rate of Heart Failure (HF) hospitalizations events for both Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB Heart Failure with reduced Ejection Fraction (HFrEF) patients | through study completion, maximum 5 years
  Heart failure hospitalizations were defined by ICD-9-CM (The International Classification of Diseases, 9th Revision, Clinical Modification) and ICD-10-CM (International Classification of Diseases, 10th Revision, Clinical Modifier) codes for HF listed within the primary diagnoses associated with a hospitalization that occurred during the follow-up period.

SECONDARY OUTCOMES:
Rate of HF hospitalizations events for both Truly naive sacubitril/valsartan HFrEF patients and Truly naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  Heart failure hospitalizations were defined by ICD-9-CM (The International Classification of Diseases, 9th Revision, Clinical Modification) and ICD-10-CM (International Classification of Diseases, 10th Revision, Clinical Modifier) codes for HF listed within the primary diagnoses associated with a hospitalization that occurred during the follow-up period.
Time to first HF hospitalization for both Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  Heart failure hospitalizations were defined by ICD-9-CM (The International Classification of Diseases, 9th Revision, Clinical Modification) and ICD-10-CM (International Classification of Diseases, 10th Revision, Clinical Modifier) codes for HF listed within the primary diagnoses associated with a hospitalization that occurred during the follow-up period.
Rate of HF hospitalizations or Emergency room (ER) visits for both Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  HF ER visits were defined by ICD-9-CM and ICD-10-CM codes for HF listed within the primary diagnoses associated with ER visits that occurred during the follow-up period.
Time to first HF hospitalization or HF ER visit for both Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  HF ER visits were defined by ICD-9-CM and ICD-10-CM codes for HF listed within the primary diagnoses associated with ER visits that occurred during the follow-up period.
Rate of all-cause hospitalizations events between Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  All-cause hospitalizations were defined as any hospitalization that occurred during the follow-up period.
Time to first all-cause hospitalizations events between Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  All-cause hospitalizations were defined as any hospitalization that occurred during the follow-up period.
Rates of cardiovascular hospitalization events between Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients | through study completion, maximum 5 years
  The rate of cardiovascular hospitalization events between Naive sacubitril/valsartan HFrEF patients and Naive ACEi/ARB HFrEF patients was reported

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CLCZ696B2036 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17872